CLINICAL TRIAL: NCT04159961
Title: A Randomized, Open-label, Parallel Design Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetic of DWJ211 in Healthy Volunteers
Brief Title: Pharmacokinetics and Safety, Tolerability of DWJ211in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWJ211101
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GroupA (Experimental): Inject the Drug into submental fat and abdominal fat via subcutaneous
  Interventions: Drug: DWJ211
- GroupB (Experimental): Inject the Drug into submental fat and abdominal fat via subcutaneous
  Interventions: Drug: DWJ211
- GroupC (Experimental): Inject the Drug into submental fat and abdominal fat via subcutaneous
  Interventions: Drug: DWJ211

INTERVENTIONS:
Drug: DWJ211 — Inject the Drug into submental fat and abdominal fat via subcutaneous

SUMMARY:
This is a randomized, open-label, parallel design Phase I clinical trial to evaluate the safety/tolerability and pharmacokinetic of DWJ211 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged between 19 and 65 at screening
* Those whose BMI is less than 40kg/m2
* Subject who will agree with the no treatment(liposuction or surgery, obesity treatment)
* Those who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* History of any intervention to treat Submental fat or abdominal fat
* History or current symptoms of dysphagia
* History of trauma associated with the chin or neck or abdominal areas that in the judgement of the investigator may affect evaluation of safety or efficacy of treatment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Cmax | 0, 5, 10, 15, 30, 45min, 1, 1.5, 2, 4, 6, 8, 12, 16, 24h
  Maximum concentration of DWJ211
Tmax | 0, 5, 10, 15, 30, 45min, 1, 1.5, 2, 4, 6, 8, 12, 16, 24h
  Time of maximum concentration
AUCt | 0, 5, 10, 15, 30, 45min, 1, 1.5, 2, 4, 6, 8, 12, 16, 24h
  Area under the drug concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No